CLINICAL TRIAL: NCT03899857
Title: Pembrolizumab for Newly Diagnosed Glioblastoma: a Prospective, Open-label, Single-arm, Multicenter Phase II Study
Brief Title: Pembrolizumab for Newly Diagnosed Glioblastoma
Acronym: PERGOLA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERGOLA
Record Dates: First submitted 2019-03-06; First posted 2019-04-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Newly Diagnosed Glioblastoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Temozolomide-based radiochemotherapy (TMZ/RT=>TMZ) represents the standard of care for patients with newly diagnosed glioblastoma. In this study, pembrolizumab will be administered (200 mg every 3 weeks) in addition to TMZ/RT=>TMZ.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be added to standard of care

SUMMARY:
The study explores the addition of pembrolizumab to temozolomide-based radiotherapy in patients with newly diagnosed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided written informed consent prior to any study-related procedure.
* Newly diagnosed glioblastoma or gliosarcoma as confirmed by local histopathology
* The patient is at least 18 years of age on day of signing informed consent
* Absence of isocitrate dehydrogenase (IDH)1 R132H mutation by immunohistochemistry
* A maximum dose of 4 mg/day dexamethasone or equivalent doses for other corticosteroids, which has been stable or decreased for ≥5 days prior to start of radiotherapy
* Patient who are treated with anticoagulants are on a stable dose for at least two weeks prior to start of radiotherapy (RT)
* The patient is male or a non-pregnant, non-lactating female
* Females of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test within 2 weeks prior to receiving the first dose of study medication. Females must practice strict birth control using two different methods (e.g. oral contraceptives in combination with barrier protection) to prevent pregnancy for the duration of the study through 120 days after the last dose of study medication. Males will be advised to use barrier protection starting with the first dose of study therapy through 120 days after the last dose of study therapy)
* The patient has a life expectancy of at least 3 months
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* The patient shows adequate organ functions as assessed by the following laboratory values within 2 weeks prior to first dose of study medication:

  * Adequate renal function determined by serum creatinine and urea < 2 times the upper limit of normal
  * Adequate liver function with alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (AP) < 3 times the upper limit of normal, and bilirubin value < 2.5 mg/dL
  * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) within therapeutic limits (according to the medical standard at the institution)
  * Hemoglobin > 9 g/dL
  * Platelet count > 100 x 10^9/L
  * White blood count (WBC) > 3 x 10^9/L
  * Absolute neutrophil count (ANC) > 1.5 x 10^9/L
* Patient is able to undergo Gd MRI.

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to temozolomide (TMZ) or pembrolizumab,
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Any known IDH mutation if tested
* Has a diagnosis of immunodeficiency
* Human immunodeficiency virus (HIV), hepatitis C virus (HBV) or hepatitis C virus (HCV) infection
* Has a history of active tuberculosis (Bacillus Tuberculosis)
* Clinically relevant acute viral, bacterial, or fungal infection
* History of a second independent malignant disorder during the last three years except non-melanoma skin cancer, in situ cervical cancer, treated superficial bladder cancer or cured, early-stage prostate cancer in a patient with prostate-specific antigen (PSA) level less than upper normal limit
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, long-term use of corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, or anti-PD-L2 agent
* Prior radiotherapy to the brain or interstitial brachytherapy
* Prior chemotherapy for a brain tumor
* Intraoperative placement of carmustine wafers (Gliadel®)
* Prior therapy with immune checkpoint inhibitors or vaccination therapy against the tumor
* Concurrent administration of any antitumor therapy other than TMZ/RT=>TMZ
* Clinically relevant psychiatric disorders/legal incapacity or a limited legal capacity
* Has received a live vaccine within 30 days of planned start of study therapy
* Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Has psychiatric or substance abuse disorders including extensive use of alcohol that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 12 months | At 12 months
  To explore whether the addition of pembrolizumab to standard temozolomide-based radiochemotherapy improves the outcome of newly diagnosed glioblastoma or gliosarcoma patients, determined by the overall survival rate at 12 months

SECONDARY OUTCOMES:
Response rates using (i)RANO (immunotherapy response assessment in neuro-oncology) criteria | From the inclusion in the study until the end of follow-up (up to approximately 36 months)
Progression-free survival (PFS) at 6 and 12 months | At 6 and 12 months
Time to treatment failure (TTF) | From the inclusion in the study until the end of follow-up (up to approximately 36 months)
Health-related Quality of life (HRQol) | From the inclusion in the study until the end of follow-up (up to approximately 36 months)
  HRQoL will be assessed with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) version 3. Scoring: 0 to 100. Higher scores mean a better level of functioning.
Correlation of programmed cell death (PD-1) ligand 1 (PD-L1) expression levels with response to treatment and outcome | From the inclusion in the study until the end of follow-up (up to approximately 36 months)
  Expression levels of PD-L1 will be determined in the tumor tissue and correlated with response as determined by MRI and progression-free as well as overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Roth, MD, Principal Investigator — University of Zurich
Locations (3):
- Switzerland (3):
  - University Hospital Bern / Inselspital, Bern
  - University Hospital Lausanne, CHUV, Lausanne
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No